CLINICAL TRIAL: NCT00210340
Title: A Phase I Study of Intrathecal Rituximab in Patients With Lymphomatous Meningitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG24
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma, B Cell
MeSH Terms: conditions — Lymphoma, B-Cell

INTERVENTIONS:
Drug: intrathecal rituximab

SUMMARY:
The purpose of this study is to define the safety profile of rituximab given intrathecally in lymphomatous meningitis related to CD20+ non-Hodgkin's lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Lymphomatous meningitis documented by positive CSF cytology in either newly diagnosed, relapsed or refractory primary CNS or systemic NHL
2. Pathologically diagnosed CD20-positive NHL
3. Age ≥ 18 years
4. ECOG Performance Status 0 - 2 (See Appendix A)
5. Life expectancy of at least 1 month
6. Informed consent must be given according to national/local regulations before enrollment (See Appendix B)
7. Patients may have had prior CNS irradiation, intrathecal methotrexate, cytarabine or thiotepa for treatment of lymphomatous meningitis but these treatments must have completed at least two weeks before the study enrollment and the patients must have recovered from any reversible toxicity caused by prior treatments
8. Concurrent systemic chemotherapy is allowed with the exception of high-dose methotrexate (>500 mg/m2/day), high-dose cytarabine (>2 g/m2/day), high-dose thiotepa (>300 mg/m2/day) or investigational agents
9. No concurrent intrathecal chemotherapy other than rituximab
10. No severe impairment of bone marrow function (ANC >1.5x109/L, PLT >50x109/L), unless due to proven lymphoma involvement
11. No major impairment of renal function (serum creatinine < 1,5 x upper normal) or liver function (ASAT/ALAT < 2,5 upper normal, total bilirubin <2,5x upper normal), unless due to proven lymphoma involvement
12. No evidence of active opportunistic infections
13. No HIV infection
14. No pregnant or lactating status
15. Appropriate contraceptive method in women of childbearing potential or men
16. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
17. Absence of a obstructive hydrocephalus or compartimentalization of CSF flow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety profile of rituximab given intrathecally

SECONDARY OUTCOMES:
preliminary evaluation of the antitumor activity of i.t. rituximab
collection of CSF samples devoted to ancillary biological studies
pharmacokinetics of different dose levels of intrathecal rituximab

CONTACTS AND LOCATIONS:
Overall Officials: Annarita Conconi, MD, Study Chair — International Extranodal Lymphoma Study Group/Hematology Division. University Amedeo Avogadro. Novara; Andres JM Ferreri, MD, Study Chair — Radiochemotherapy San Raffaele Hospital. Milan

REFERENCES:
- See also: Click here for more information about this study: phase I study of intrathecal rituximab in patients with lymphomatous meningitis — http://www.ielsg.org